CLINICAL TRIAL: NCT06062459
Title: Synergistic Benefits of Motor Control Exercises and Balance Training in Sacroiliac Joint Dysfunction: A Randomized Controlled Trial
Brief Title: Synergistic Benefits of MCE and BT in Sacroiliac Joint Dysfunction: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IE/IIMS&R/2022/87
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Sacroiliac Joint Dysfunction
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): MCE Group
  Interventions: Other: Motor Control Exercise; Other: Control Group
- Group B (Experimental): BT Group
  Interventions: Other: Balance Training; Other: Control Group
- Group C (Experimental): Combined MCE & BT Group
  Interventions: Other: Motor Control Exercise; Other: Balance Training; Other: Control Group
- Group D (Other): Control Group
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Motor Control Exercise — Motor control exercises focusing on the activation and control of deep spinal muscles
  Arms: Group A; Group C
Other: Balance Training — Balance training exercises on to enhance proprioception and stability
  Arms: Group B; Group C
Other: Control Group — Participants received hot pack and stretching exercise

SUMMARY:
This research aimed to ascertain the combined and individual efficacies of MCE and BT in alleviating SIJD symptoms.

DETAILED DESCRIPTION:
The study will be based on a four-arm parallel group randomized control design. one hundred and twenty participants with SIJD will be recruited from the Physiotherapy department, at Integral University, India. Study objectives and procedure will be properly explained and written informed consent will be obtained at the beginning of the study. All the participants will be randomly divided into four groups A, B, C, and D. Experimental group A will be receiving the hot pack, Stretching exercise, and MCE intervention, group B will receive the hot pack, Stretching exercise, and BT exercise and Group C will be receiving the hot pack, Stretching exercise, and MCE & BT intervention, control group D will receive the hot pack, Stretching exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age-30-60 Years
* sacroiliac joint pain (>3 months)
* Presence of pain exacerbated as a result of bending laterally or backward
* Positive results on at least 2 of the pain-provocation tests [FABER, Posterior shear and Gaenslen pain provocation tests) and one of the motion palpation tests (ie, Gillet and forward flexion tests)

Exclusion Criteria:

* past or current history of surgery or major trauma to spine, pelvis, lower limb, chest or abdomen in the past 12 months
* lower extremity musculoskeletal disorders; known localized spinal pathology
* known congenital anomalies of hip, pelvis or spine that limits mobility
* known systematic arthropathy, neuropathy or metabolic disorder
* Presence of other causes of LBP such as lumbar discopathy and spinal stenosis discovered via clinical examination and MRI scanning
* pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 Weeks
  The pain intensity was assessed Using a numeric pain rating scale (NPRS), It's a 11 point scale, where zero indicates no pain and 10 indicates severe pain
Functional disability | 6 Weeks
  Functional limitation was assessed by using Oswestry disability Index questionnaire Each section is scored on a 0-5 scale, 5 representing the greatest disability.
self-reported measure of health | 6 Weeks
  It comprises 36 questions that cover eight domains of health

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, Principal Investigator — Najran University
Locations (2):
- Integral University Hospital, Lucknow, Uttar Pardesh, India
- Hashim Ahmed, Najrān, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No